CLINICAL TRIAL: NCT05321485
Title: The Effect of MedicijnWijs on Adherence to Azathioprine Therapy in Adolescents With IBD
Acronym: MEDICATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, dr. L.J.J. (Luc) Derijks, L.J.J. (Luc) Derijks, PharmD, PhD, hospital pharmacist-clinical pharmacologist, Maxima Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-MMC-029
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Adherence; Azathioprine; Knowledge; App; Phone; Education
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MedicijnWijs (Experimental): All participants will undergo the same intervention of using MedicijnWijs, and they will serve as their own control.
  Interventions: Other: MedicijnWijs

INTERVENTIONS:
Other: MedicijnWijs — The mobile phone app MedicijnWijs will guide the participants with their azathioprine therapy during 6 weeks. Information about azathioprine is given as well as general information about IBD, specified to disease modality (Crohn's Disease and Ulcerative Colitis). Contact details of the patient's pharmacy are listed, questions about the patient's symptoms are asked, and push notifications are added to remind the patients to take their medication.
  At the beginning of the 6-weeks guidance, two validated questionnaires that are translated and validated in Dutch will have to be filled in: the MARS-5 and the IBD-KID2. After 6 weeks, the participants have to fill out the same questionnaires again to assess potential changes in the scores compared to baseline. Also, a number of questions will be asked to assess the ease of use of MedicijnWijs.

SUMMARY:
Medication non-adherence is an existing problem in patients with inflammatory bowel diseases (IBD). Adherence rates are especially low in children and adolescents. Good medication adherence is key in achieving lower disease activity and longer periods of remission. Previous research has shown education can increase medication adherence. MedicijnWijs is a mobile phone app containing a module concerning a 6-weeks guidance with azathioprine therapy. It provides information about IBD and azathioprine. In this multicenter before-and-after study, the aim is to assess the effect of MedicijnWijs on the adherence to azathioprine therapy in adolescents with IBD. This is done using two validated questionnaires that are translated to Dutch: the Medication Adherence Report Scale-5 (MARS-5), which tests the participants' adherence to azathioprine therapy, and the Inflammatory Bowel Disease Knowledge Inventory Device 2 (IBD-KID2), which tests the participants' knowledge about IBD. These questionnaires are filled in at the beginning of the study period and after 6 weeks of using MedicijnWijs. This way a change in both scores can be assessed. The investigators hypothesize that MedicijnWijs will help increase the adherence to azathioprine therapy in adolescents with IBD.

DETAILED DESCRIPTION:
Rationale: medication non-adherence is an existing problem in patients with inflammatory bowel diseases (IBD). Adherence rates are especially low in children and adolescents. Good medication adherence is key in achieving lower disease activity and longer periods of remission. Previous research has shown education can increase medication adherence. MedicijnWijs is a mobile phone app containing a module concerning a 6-weeks guidance with azathioprine therapy. The aim of this study is to assess the effect of MedicijnWijs on the adherence to azathioprine therapy in adolescents with IBD. The investigators hypothesize that MedicijnWijs will help increase the adherence to azathioprine therapy in adolescents with IBD.

Objective: with this study, the effect of the mobile phone app MedicijnWijs on adherence to azathioprine therapy will be assessed. In addition, the effect on knowledge about IBD and the ease of use of MedicijnWijs will be studied as well.

Study design: this study is a multicenter before-and-after study. Study population: the study population are adolescents aged 12 up to and including 17 years old. All participants are diagnosed with IBD and are treated with azathioprine. This multicenter study will be conducted in Máxima Medical Center in Veldhoven, Catharina Hospital in Eindhoven, and Zuyderland Medical Center in Sittard-Geleen/Heerlen, The Netherlands.

Intervention: the participants will use the mobile phone app MedicijnWijs for 6 weeks. In this app, information about IBD and azathioprine is provided. Participants also receive questions about their symptoms through the app. Moreover, at the beginning of the study the participants have to fill in two validated questionnaires that are translated to Dutch in the app: the Medication Adherence Report Scale-5 (MARS-5), which tests the participants' adherence to azathioprine therapy, and the Inflammatory Bowel Disease Knowledge Inventory Device 2 (IBD-KID2), which tests the participants' knowledge about IBD. After 6 weeks, the participants have to fill out the same questionnaires again to assess potential changes in the scores compared to baseline. Also, a number of questions will be asked to assess the ease of use of MedicijnWijs.

Main study parameters/endpoints: the main endpoint is change in adherence to azathioprine therapy measured as a change in MARS-5 score. In addition, the secondary endpoint change in knowledge about IBD measured as a change in IBD-KID2 score will be studied as well. The results of the secondary endpoint ease of use of MedicijnWijs will be presented descriptively.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: there are no risks associated with participation to this study as participants only have to use a mobile phone app and fill in two short questionnaires. MedicijnWijs has to be used for 6 weeks. The time burden per day varies from 0 to 10 minutes. The IBD treatment of the participants will not change, and participants will visit their doctors as frequently as usual. Only an additional introductory talk will be necessary, which will be scheduled during a regular outpatient clinic visit. No physical examinations, blood tests, or other tests will be done during this study apart from routine care of IBD.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12 up to and including 17 years old
* Condition: IBD (Crohn's Disease and Ulcerative Colitis)
* Treatment: azathioprine

Exclusion Criteria:

- Inability to use MedicijnWijs due to either low cognitive skills or the unavailability of a phone or other technical device to use the app on

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-09-16 (Estimated); Study Completion 2022-09-16 (Estimated)

PRIMARY OUTCOMES:
Change in adherence to azathioprine therapy | 6 weeks
  Measured as the change in Medication Adherence Report Scale-5 (MARS-5) score compared to baseline. The MARS-5 score at the start and end of the study can range from 5 to 25 points. The higher the score, the better the adherence to azathioprine therapy. The difference in MARS-5 score compared to baseline will be assessed.

SECONDARY OUTCOMES:
Change in knowledge about IBD | 6 weeks
  Measured as the change in Inflammatory Bowel Disease-Knowledge Inventory Device 2 (IBD-KID2) score compared to baseline. The IBD-KID2 score at the start and end of the study can range from 0 to 15 points. The higher the score, the higher the knowledge about IBD. The difference in IBD-KID2 score compared to baseline will be assessed.
Ease of use of MedicijnWijs assessed by a questionnaire | At the end of 6 weeks
  Assessed by separate questions

CONTACTS AND LOCATIONS:
Overall Officials: Luc JJ Derijks, PharmD, PhD, Principal Investigator — Maxima Medical Center
Locations (3):
- Netherlands (3):
  - Catharina Hospital, Eindhoven, North Brabant
  - Zuyderland Medisch Centrum, Heerlen, North Brabant
  - Maxima Medical Center, Veldhoven, North Brabant

IPD SHARING:
Plan to Share IPD: No